CLINICAL TRIAL: NCT06406218
Title: The Impact of Phase I Cardiac Rehabilitation on the Prognosis of Acute Myocardial Infarction (AMI) Patients After Percutaneous Coronary Intervention (PCI): A Single-Center, Randomized Controlled Study
Brief Title: The Impact of Phase I Cardiac Rehabilitation on the Prognosis of AMI Patients After PCI
Acronym: AID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Han Yaling, MD (Other)
Responsible Party: Sponsor-Investigator, Han Yaling, MD, Chief Physician, Shenyang Northern Hospital
Organization: Shenyang Northern Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AID
Record Dates: First submitted 2024-04-29; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Acute Myocardial Infarction; Phase I Cardiac Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase I Cardiac Rehabilitation Exercise Training (Experimental)
  Interventions: Behavioral: Phase I Cardiac Rehabilitation Exercise Training
- Guideline control (No Intervention): During hospitalization, patients assigned to the guideline control only receive routine medication treatment according to the guidelines, without any exercise intervention or education.

INTERVENTIONS:
Behavioral: Phase I Cardiac Rehabilitation Exercise Training — A) In the morning, take a supine position and perform straight leg raises with each leg individually, lifting to a height of 30° and holding for 3-5 seconds. Raise both arms to the side of the head to a 90° angle and hold for 5-10 seconds. Inhale deeply when exerting force and exhale slowly when lowering. Alternate between leg lifts and arm raises, performing 5 sets per session. Adjust intensity based on individual condition and may be repeated. In the afternoon, sit beside the bed for 5 minutes. B) After transitioning to secondary care according to the patient's condition, stand beside the bed for 5 minutes in the morning; in the afternoon, march in place beside the bed for 5 minutes. C) Walk beside the bed for 10 minutes per session, twice a day. D) Move around and doing activities under supervision inside the ward, 10 minutes per session, twice a day.
  Spend approximately one day at each level, gradually progressing the exercise to the patient's tolerance level.
  Arms: Phase I Cardiac Rehabilitation Exercise Training

SUMMARY:
Previous research has confirmed that patients undergoing percutaneous coronary intervention (PCI) can benefit from cardiac rehabilitation programs. However, there is a paucity of studies on Phase I cardiac rehabilitation commenced within three days following PCI in patients with acute myocardial infarction (AMI). Consequently, the objective of the study is to demonstrate whether Phase I cardiac rehabilitation can improve the prognosis at 12 months when compared with the control group. The primary endpoint is the Seattle Angina Questionnaire (SAQ) score at 12 months for the patients. The principal hypothesis of the study is that Phase I cardiac rehabilitation will improve the long-term prognosis for AMI patients at 12 months after PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AMI (including STEMI and NSTEMI) who were treated in the CCU (Coronary Care Unit) for more than 12 hours after emergency PCI;
2. Patients who are expected to meet the discharge criteria without the need for repeat PCI during the current hospital stay after PCI;
3. No chest pain episodes within 8 hours, with no recurrence of myocardial infarction; remained hemodynamically stable;
4. No further increase in serum levels of cardiac biomarkers such as Creatine Kinase -MB (CK-MB) and cardiac troponins (cTn).

Exclusion Criteria:

1. Patients with Killip class III or higher, or symptoms and signs of acute pulmonary edema and respiratory distress;
2. Malignant arrhythmias that cause hemodynamic instability and potentially life-threatening conditions;
3. Mechanical lesions such as ventricular wall rupture, valve or tendon rupture;
4. Patients who have not yet been weaned off ECMO, IABP, temporary pacemakers, CRRT;
5. Patients with liver or kidney dysfunction (transaminase exceeded three times the upper limit of normal; EGFR<30 ml/(min·1.73m^2)) or advanced malignant tumors;
6. Patients who cannot undergo exercise rehabilitation due to orthopedic or psychiatric diseases;
7. Patients with language impairment;
8. Patients currently undergoing systematic training or participating in other clinical trials without reaching the primary endpoint collection time;
9. Researchers believe that patients are not suitable for participation in this study or have not obtained an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Seattle Angina Questionnaire (SAQ) | 6-month and 12-month
  Seattle Angina Questionnaire Score (from 0 to 500) higher scores mean a better outcome.
  The assessment consists of five specific dimensions, with each dimension scored on a scale ranging from 0 to 100.
  1. Degree of physical activity limitation.
  2. Stable angina status.
  3. Frequency of angina attacks.
  4. Satisfaction with treatment.
  5. Level of disease awareness.

SECONDARY OUTCOMES:
6 minutes walking distance | 6-month and 12-month
Left ventricular ejection fraction | 6-month
  The percentage of the left ventricular stroke volume relative to the left ventricular end-diastolic volume(%).
MACCE | 12-month
  All-cause death, myocardial infarction, stroke, revascularization again

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Ling Han, PhD, Principal Investigator — Department of Cardiology, General Hospital of Northern Theater Command, Shenyang 110016, China
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No